CLINICAL TRIAL: NCT01302535
Title: The Impact of Yoga on Blood Pressure and Quality of Life in Patients With Hypertension - a Randomised Controlled Trial in Primary Health Care
Brief Title: The Impact of Yoga on Blood Pressure and Quality of Life in Patients With Hypertension
Acronym: YHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Moa Wolff, General practitioner, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/728
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension
Keywords: Yoga; Hypertension; Quality of Life; Primary Health Care
MeSH Terms: conditions — Hypertension | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga group with supervision/trainer (Active Comparator)
  Interventions: Other: Yoga group with supervision (trainer)
- Yoga at home (Active Comparator)
  Interventions: Other: Yoga at home
- Control (No Intervention): No changes will be made for the participants in the control group, but they will undergo the same measurements and evaluations as the intervention groups.

INTERVENTIONS:
Other: Yoga group with supervision (trainer) — The Yoga-with-trainer group will meet once a week (60 minutes) to practice yoga with a yoga instructor. The participants will be encouraged to practice yoga between the yoga classes at home for 30 minutes a day.
  Arms: Yoga group with supervision/trainer
Other: Yoga at home — The participants in the Yoga-at-home group will get a private doctor appointment (20 minutes) where they get instructions for two yoga exercises which they are encouraged to perform at home 15 minutes a day.
  Arms: Yoga at home

SUMMARY:
The purpose of this study is to determine the effects of yoga on blood pressure and quality of life in patients in primary health care diagnosed with hypertension within the last year. Another purpose is to examine whether the possible effect on blood pressure differs if patients practice yoga in a group lead by a yoga-trainer or receive a few yoga-exercises from their doctor to be practiced individually at home.

DETAILED DESCRIPTION:
Hypertension is one of the most common diseases in the industrialized world. In Sweden alone approximately 1.8 million persons, 25% of the adult population, have hypertension. Hypertension is a common diagnosis in primary health care and the costs of investigating and treating hypertension and its consequences are considerable. We know that stress can affect blood pressure, but it is hard to measure and control.

Previous studies have separately shown that yoga can reduce levels of cortisol in saliva and lower blood pressure. However, few studies have investigated the effects of yoga on hypertension and we lack information about the possibility of using yoga in primary health care to reduce hypertension.

If yoga can be used to complement antihypertensive medicines, it could reduce medicine intake and thereby possibly reduce side effects and lower medicine costs. It is to be hoped that patients will also experience a higher quality of life if they perform yoga on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hypertension since at least one year.
* Blood pressure 120/80-160/100 mmHg at the last blood pressure control by doctor or nurse.

Exclusion Criteria:

* Blood pressure >180 systolic and/or >110 diastolic by the initial control in the study.
* Blood pressure <120 systolic by the initial control in the study.
* Medical adjustments regarding hypertension within 4 weeks prior to begin of study.
* Expected inability to understand instructions about yoga exercises (e.g dementia and mental retardation) or physical or psychical inability to carry out yoga exercises (e.g severe physical or psychical handicap).
* Need for interpreter. Linguistic/language difficulties
* Older than 80 years

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hypertension | 12 weeks
  At the beginning of the study, all subjects will undergo a standardized blood pressure test with an hypertension monitor. After 12 weeks, all subjects in the intervention and control groups will again be requested to attend a blood pressure testing session. Blood samples will also be collected and analysed in the beginning and at the end of the study. Some blood samples will be preserved for future analysis.

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  At the beginning of the study, all subjects will be requested to fill in a questionnaire about their quality of life (WHOQOL-BREF). After 12 weeks all subjects in the intervention and control groups will fill in the quality of life-form for a second time.

CONTACTS AND LOCATIONS:
Overall Officials: Moa Wolff, MD, Principal Investigator — Center for Primary Health Care Research, Lunds University
Locations (1):
- Center for Primary Health Care Research, Lunds University, Malmo, Sweden

REFERENCES:
- [Derived] Wolff M, Memon AA, Chalmers JP, Sundquist K, Midlov P. Yoga's effect on inflammatory biomarkers and metabolic risk factors in a high risk population - a controlled trial in primary care. BMC Cardiovasc Disord. 2015 Aug 19;15:91. doi: 10.1186/s12872-015-0086-1. PMID 26286137
- [Derived] Wolff M, Sundquist K, Larsson Lonn S, Midlov P. Impact of yoga on blood pressure and quality of life in patients with hypertension - a controlled trial in primary care, matched for systolic blood pressure. BMC Cardiovasc Disord. 2013 Dec 7;13:111. doi: 10.1186/1471-2261-13-111. PMID 24314119